CLINICAL TRIAL: NCT07180680
Title: Preliminary Results of Laparoscopic Assisted Transanal Proximal Rectosigmoidectomy Combined With Malone Antegrade Continence Enema for the Management of Intractable Functional Constipation in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelmaboud, Assistant professor of pediatric surgery, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PedSurg-38Med.Research.0000038
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Functional Constipation in Children
Keywords: Intractable functional constipation; laparoscopic rectosigmoidectomy; pediatric; quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children diagnosed with IFC (Active Comparator): . Each participant underwent LATPRS combined with a Malone Antegrade continence enema (MACE)
  Interventions: Procedure: laparoscopic assisted transanal proximal rectosigmoidectomy

INTERVENTIONS:
Procedure: laparoscopic assisted transanal proximal rectosigmoidectomy — using laparoscopy for such procedure in children is unique for this study

SUMMARY:
Technique for surgical management of intractable functional constipation

DETAILED DESCRIPTION:
Background: Intractable functional constipation (IFC) in children poses a significant clinical challenge when standard medical interventions are unsuccessful. The laparoscopic-assisted transanal proximal rectosigmoidectomy (LATPRS) procedure is a surgical option that combines the precision of laparoscopic techniques with the functional benefits of transanal dissection.

Patients and methods: A prospective trial was conducted at Al-Azhar pediatric surgery departments from January 2022 to January 2025, with a focus on children diagnosed with IFC. Each participant underwent LATPRS combined with a Malone Antegrade continence enema (MACE). The comprehensive data collection process included patient demographics, surgical details, postoperative recovery, complications, and functional outcomes. These data were recorded and subsequently analysed. Furthermore, a validated symptom severity (SS) scoring system and the Pediatric Quality of Life Inventory (PedsQoL) were employed to assess outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged four years or older with intractable functional constipation
2. Documented BMP failure, defined as persistent fecal impaction, chronic dependence on laxatives, or intolerance to enemas despite prolonged conservative therapy.

Exclusion Criteria:

1. Patients with a history of abdominal surgery or
2. Identifiable organic causes for constipation and soiling (e.g., Hirschsprung's disease, anorectal malformations, or metabolic disorders) .

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
soiling | 3 years
  Number of soiling episodes in pre-operative and post-operative period. Soiling refers to the inadvertent passage of fecal material into inappropriate places, such as underwear or other clothing.

SECONDARY OUTCOMES:
symptoms severity score | 3 years
  The total symptoms severity score ranged from 0, indicating the best outcome, to 65, indicating the worst outcome. These scores comprised individual assessments in the following areas: soiling problems (range = 0--10); delay in defecation (range = 0--10); difficulty and pain associated with stool passage (range = 0--5); intensity of laxative treatment (range = 0--10); child's general health (range = 0--5); behavior related to bowel problems (range = 0--5); overall improvement of symptoms (range = 0--12); and amount of stool detected during abdominal examination (range = 0--8). A score range of 0-21 is classified as mild and considered "well." In contrast, a score range of 22-43 is categorized as moderate, indicating noticeable bowel dysfunction that requires ongoing management. A score ranging from 44-65 is classified as severe, with significant debilitating symptoms indicative of intractable cases
The Pediatric Quality of Life Inventory (The PedsQoL™ questionnaires) | 3 years
  The tool initially created by James W. Varni and colleagues [16], which has received prior validation from the World Health Organization, was employed to evaluate QoL. This is a practical and validated modular tool for assessing health-related quality of life (HRQOL) in children aged 4-18 years (10). The scale evaluates the fundamental aspects of physical, emotional, social, and school functioning in children. The PedsQoL total score ranges from 0 to 92. A score between 0 and 30 is regarded as having a mild impact, indicating good quality of life. In contrast, a score between 31 and 61 suggests a moderate impact with some limitations in physical, emotional, or social functioning. A score from 62 to 92 is considered to have a severe impact, reflecting a significant compromise in quality of life, with notable distress or disability

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelmaboud, assistant professor, Principal Investigator — Faculty of medicine- Al-Azhar University Hospitals
Locations (1):
- pediatric surgery departments- Al-Azhar University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided